CLINICAL TRIAL: NCT04687176
Title: Frontline Oral Arsenic Trioxide-based Induction in Newly Diagnosed Acute Promyelocytic Leukaemia
Brief Title: Frontline Oral Arsenic Trioxide for APL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL003
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-09

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia; Oral Arsenic Trioxide; Chemotherapy-free
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral arsenic trioxide, all-trans-retinoic acid, ascorbic acid (AAA) (Experimental): Induction: Oral arsenic trioxide 10mg daily (0.16mg/kg/day in patients < 18 years-old, all-trans retinoic acid (ATRA) [45mg/m^2 (25mg/m^2 per day in patients < 18 years-old) in 2 divided doses) and ascorbic acid 1g daily (15mg/kg/day in patients < 18 years-old) for 42 days Consolidation: Oral arsenic trioxide daily, ATRA, and ascorbic acid daily for 14 days every 28 days for 2 cycles.
  Maintenance: Oral arsenic trioxide, ATRA and ascorbic acid daily for 2 weeks every 8 weeks for a total of 2 years (i.e. for 12 cycles in total).
  Interventions: Drug: Oral Arsenic Trioxide Formulation

INTERVENTIONS:
Drug: Oral Arsenic Trioxide Formulation — Patients will be recruited to oral arsenic trioxide, all-trans-retinoic acid, ascorbic acid (AAA) based-induction for 42 days. Daunorubicin or idarubicin will only be used during induction in patients <65 with presenting white blood cell count (WBC) ≥ 10 x 10^9/L. In patients not receiving daunorubicin, hydroxyurea if WBC ≥ 5 x 10^9/L within the first 14 days of induction. A reassessment bone marrow aspirate will be performed on day 28 of induction for assessment of morphologic remission.
  Four weeks after the completion of induction phase, all patients, regardless of initial WBC, will receive two cycles of chemotherapy-free AAA consolidation (14 days every 28 days).
  Four weeks after completion of consolidation, all patients will receive 12 cycles of chemotherapy-free AAA maintenance (14 days every 8 week).
  Other Names: ARSENOL

SUMMARY:
The investigators have formulated an oral preparation of arsenic trioxide (oral-ATO), and shown that it is efficacious for APL in R1, inducing CR2 in more than 90% of patients [8,9]. Furthermore, in an effort to prevent relapse, the investigators have moved oral-ATO forward to the maintenance of CR1. This strategy results in favorable overall-survival (OS) and leukemia-free-survival (LFS) [10], implying that prolonged treatment with oral-ATO may prevent relapses.

Current protocols have incorporated i.v.-ATO in the treatment of newly-diagnosed APL [11-15]. For regimens comprising oral-ATO, ATRA and chemotherapy, 5-year OS in excess of 90% is achieved [11-15].

The investigators have also published long-term data showing the use of oral-ATO is highly effective and safe in the relapsed and frontline settings [16,17].

In this study, the investigators evaluate the use of oral-ATO and ATRA based induction regimens in newly diagnosed patients with APL with no of minimal chemotherapy in a prospective multicentre phase 2 study.

DETAILED DESCRIPTION:
After initial eligibility screening, patients will be recruited to oral arsenic trioxide, all-trans-retinoic acid, ascorbic acid (AAA) based-induction for 42 days. Daunorubicin or idarubicin will only be used during induction in patients <65 with presenting white blood cell count (WBC) ≥ 10 x 10^9/L. In patients not receiving daunorubicin, hydroxyurea if WBC ≥ 5 x 10^9/L within the first 14 days of induction. Molecular monitoring monitoring with RQ-PCR or ddPCR for PML-RARA will be performed weekly during induction. A reassessment bone marrow aspirate will be performed on day 28 of induction for assessment of morphologic remission.

Four weeks after the completion of induction phase, all patients, regardless of initial WBC, will receive two cycles of chemotherapy-free AAA consolidation (14 days every 28 days).

Four weeks after completion of consolidation, all patients will receive 12 cycles of chemotherapy-free AAA maintenance (14 days every 8 week).

Molecular monitoring monitoring with RQ-PCR or ddPCR for PML-RARA will be performed during every 4 weeks during consolidation, every 8 weeks during maintenance, and every 3 months for 24 months after completion of maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed APL with t(15;17)(q24;q21) or acute myeloid leukaemia (AML) with variant RARA translocation according to the World Health Organization (WHO) Classification 2022
2. Ability and willingness to comply with the study procedures and restrictions
3. Voluntary written informed consent

Exclusion Criteria:

1. ECOG performance score >2
2. Decompensated heart failure with left-ventricular ejection fraction of less than 40% and global hypokinesia on echocardiogram.
3. Prolonged corrected QT interval (QTc) ≥ 500ms, in the absence of electrolyte disturbances and medications known to prolong QTc
4. Significant liver function derangement (Bilirubin > 3 times upper limit normal and/or ALT > 5 times upper limit of normal)
5. Glomerular filtration rate (GRF) by Cockcroft-Gault formula or eGFR (MDRD) of less than 30mL/min in adults (aged ≥ 18) or Creatinine clearance < 50ml/min/1.73m2 in paediatric and adolescent patients (Age ≤ 17)
6. Female subject who is lactating or has positive pregnancy test result prior to the first dose of study drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 60 months
  Defined as the time (in months) from first complete morphologic remission (CR1) to morphologic or molecular relapse (event), or latest follow-up (censored).
Event-free survival (EFS) | 60 months
  Defined as the time (in months) from recruitment to treatment failure (event), morphologic or molecular relapse (event), or latest follow-up (censored).

SECONDARY OUTCOMES:
Overall survival | 60 months
  Defined as time (in months) from diagnosis to death (event) or latest follow-up (censored).
Treatment toxicities | 60 months
  Treatment toxicities by Common Toxicity Criteria for Adverse Everts (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Gill, MD, Principal Investigator — The University of Hong Kong
Locations (2):
- The University of Hong Kong, Hong Kong, Hong Kong
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tallman MS, Altman JK. How I treat acute promyelocytic leukemia. Blood. 2009 Dec 10;114(25):5126-35. doi: 10.1182/blood-2009-07-216457. PMID 19797519
- [Background] Tallman MS, Andersen JW, Schiffer CA, Appelbaum FR, Feusner JH, Woods WG, Ogden A, Weinstein H, Shepherd L, Willman C, Bloomfield CD, Rowe JM, Wiernik PH. All-trans retinoic acid in acute promyelocytic leukemia: long-term outcome and prognostic factor analysis from the North American Intergroup protocol. Blood. 2002 Dec 15;100(13):4298-302. doi: 10.1182/blood-2002-02-0632. Epub 2002 Aug 15. PMID 12393590
- [Background] Lengfelder E, Haferlach C, Saussele S, Haferlach T, Schultheis B, Schnittger S, Ludwig WD, Staib P, Aul C, Gruneisen A, Kern W, Reichle A, Serve H, Berdel WE, Braess J, Spiekermann K, Wormann B, Sauerland MC, Heinecke A, Hiddemann W, Hehlmann R, Buchner T; German AML Cooperative Group. High dose ara-C in the treatment of newly diagnosed acute promyelocytic leukemia: long-term results of the German AMLCG. Leukemia. 2009 Dec;23(12):2248-58. doi: 10.1038/leu.2009.183. Epub 2009 Sep 10. PMID 19741727
- [Background] Lo-Coco F, Avvisati G, Vignetti M, Breccia M, Gallo E, Rambaldi A, Paoloni F, Fioritoni G, Ferrara F, Specchia G, Cimino G, Diverio D, Borlenghi E, Martinelli G, Di Raimondo F, Di Bona E, Fazi P, Peta A, Bosi A, Carella AM, Fabbiano F, Pogliani EM, Petti MC, Amadori S, Mandelli F; Italian GIMEMA Cooperative Group. Front-line treatment of acute promyelocytic leukemia with AIDA induction followed by risk-adapted consolidation for adults younger than 61 years: results of the AIDA-2000 trial of the GIMEMA Group. Blood. 2010 Oct 28;116(17):3171-9. doi: 10.1182/blood-2010-03-276196. Epub 2010 Jul 19. PMID 20644121
- [Background] Kelaidi C, Chevret S, De Botton S, Raffoux E, Guerci A, Thomas X, Pigneux A, Lamy T, Rigal-Huguet F, Meyer-Monard S, Chevallier P, Maloisel F, Deconinck E, Ferrant A, Fegueux N, Ifrah N, Sanz M, Dombret H, Fenaux P, Ades L. Improved outcome of acute promyelocytic leukemia with high WBC counts over the last 15 years: the European APL Group experience. J Clin Oncol. 2009 Jun 1;27(16):2668-76. doi: 10.1200/JCO.2008.18.4119. Epub 2009 May 4. PMID 19414681
- [Background] Niu C, Yan H, Yu T, Sun HP, Liu JX, Li XS, Wu W, Zhang FQ, Chen Y, Zhou L, Li JM, Zeng XY, Yang RR, Yuan MM, Ren MY, Gu FY, Cao Q, Gu BW, Su XY, Chen GQ, Xiong SM, Zhang TD, Waxman S, Wang ZY, Chen Z, Hu J, Shen ZX, Chen SJ. Studies on treatment of acute promyelocytic leukemia with arsenic trioxide: remission induction, follow-up, and molecular monitoring in 11 newly diagnosed and 47 relapsed acute promyelocytic leukemia patients. Blood. 1999 Nov 15;94(10):3315-24. PMID 10552940
- [Background] Soignet SL, Frankel SR, Douer D, Tallman MS, Kantarjian H, Calleja E, Stone RM, Kalaycio M, Scheinberg DA, Steinherz P, Sievers EL, Coutre S, Dahlberg S, Ellison R, Warrell RP Jr. United States multicenter study of arsenic trioxide in relapsed acute promyelocytic leukemia. J Clin Oncol. 2001 Sep 15;19(18):3852-60. doi: 10.1200/JCO.2001.19.18.3852. PMID 11559723
- [Background] Au WY, Kumana CR, Kou M, Mak R, Chan GC, Lam CW, Kwong YL. Oral arsenic trioxide in the treatment of relapsed acute promyelocytic leukemia. Blood. 2003 Jul 1;102(1):407-8. doi: 10.1182/blood-2003-01-0298. No abstract available. PMID 12814916
- [Background] Au WY, Li CK, Lee V, Yuen HL, Yau J, Chan GC, Ha SY, Kwong YL. Oral arsenic trioxide for relapsed acute promyelocytic leukemia in pediatric patients. Pediatr Blood Cancer. 2012 Apr;58(4):630-2. doi: 10.1002/pbc.23306. Epub 2011 Sep 2. PMID 21898784
- [Background] Au WY, Kumana CR, Lee HK, Lin SY, Liu H, Yeung DY, Lau JS, Kwong YL. Oral arsenic trioxide-based maintenance regimens for first complete remission of acute promyelocytic leukemia: a 10-year follow-up study. Blood. 2011 Dec 15;118(25):6535-43. doi: 10.1182/blood-2011-05-354530. Epub 2011 Oct 12. PMID 21998212
- [Background] Hu J, Liu YF, Wu CF, Xu F, Shen ZX, Zhu YM, Li JM, Tang W, Zhao WL, Wu W, Sun HP, Chen QS, Chen B, Zhou GB, Zelent A, Waxman S, Wang ZY, Chen SJ, Chen Z. Long-term efficacy and safety of all-trans retinoic acid/arsenic trioxide-based therapy in newly diagnosed acute promyelocytic leukemia. Proc Natl Acad Sci U S A. 2009 Mar 3;106(9):3342-7. doi: 10.1073/pnas.0813280106. Epub 2009 Feb 18. PMID 19225113
- [Background] Iland HJ, Bradstock K, Supple SG, Catalano A, Collins M, Hertzberg M, Browett P, Grigg A, Firkin F, Hugman A, Reynolds J, Di Iulio J, Tiley C, Taylor K, Filshie R, Seldon M, Taper J, Szer J, Moore J, Bashford J, Seymour JF; Australasian Leukaemia and Lymphoma Group. All-trans-retinoic acid, idarubicin, and IV arsenic trioxide as initial therapy in acute promyelocytic leukemia (APML4). Blood. 2012 Aug 23;120(8):1570-80; quiz 1752. doi: 10.1182/blood-2012-02-410746. Epub 2012 Jun 19. PMID 22715121
- [Background] Lo-Coco F, Avvisati G, Vignetti M, Thiede C, Orlando SM, Iacobelli S, Ferrara F, Fazi P, Cicconi L, Di Bona E, Specchia G, Sica S, Divona M, Levis A, Fiedler W, Cerqui E, Breccia M, Fioritoni G, Salih HR, Cazzola M, Melillo L, Carella AM, Brandts CH, Morra E, von Lilienfeld-Toal M, Hertenstein B, Wattad M, Lubbert M, Hanel M, Schmitz N, Link H, Kropp MG, Rambaldi A, La Nasa G, Luppi M, Ciceri F, Finizio O, Venditti A, Fabbiano F, Dohner K, Sauer M, Ganser A, Amadori S, Mandelli F, Dohner H, Ehninger G, Schlenk RF, Platzbecker U; Gruppo Italiano Malattie Ematologiche dell'Adulto; German-Austrian Acute Myeloid Leukemia Study Group; Study Alliance Leukemia. Retinoic acid and arsenic trioxide for acute promyelocytic leukemia. N Engl J Med. 2013 Jul 11;369(2):111-21. doi: 10.1056/NEJMoa1300874. PMID 23841729
- [Background] Abaza Y, Kantarjian H, Garcia-Manero G, Estey E, Borthakur G, Jabbour E, Faderl S, O'Brien S, Wierda W, Pierce S, Brandt M, McCue D, Luthra R, Patel K, Kornblau S, Kadia T, Daver N, DiNardo C, Jain N, Verstovsek S, Ferrajoli A, Andreeff M, Konopleva M, Estrov Z, Foudray M, McCue D, Cortes J, Ravandi F. Long-term outcome of acute promyelocytic leukemia treated with all-trans-retinoic acid, arsenic trioxide, and gemtuzumab. Blood. 2017 Mar 9;129(10):1275-1283. doi: 10.1182/blood-2016-09-736686. Epub 2016 Dec 21. PMID 28003274
- [Background] Burnett AK, Russell NH, Hills RK, Bowen D, Kell J, Knapper S, Morgan YG, Lok J, Grech A, Jones G, Khwaja A, Friis L, McMullin MF, Hunter A, Clark RE, Grimwade D; UK National Cancer Research Institute Acute Myeloid Leukaemia Working Group. Arsenic trioxide and all-trans retinoic acid treatment for acute promyelocytic leukaemia in all risk groups (AML17): results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2015 Oct;16(13):1295-305. doi: 10.1016/S1470-2045(15)00193-X. Epub 2015 Sep 14. PMID 26384238
- [Background] Gill H, Yim R, Lee HKK, Mak V, Lin SY, Kho B, Yip SF, Lau JSM, Li W, Ip HW, Hwang YY, Chan TSY, Tse E, Au WY, Kumana CR, Kwong YL. Long-term outcome of relapsed acute promyelocytic leukemia treated with oral arsenic trioxide-based reinduction and maintenance regimens: A 15-year prospective study. Cancer. 2018 Jun 1;124(11):2316-2326. doi: 10.1002/cncr.31327. Epub 2018 Mar 26. PMID 29579321
- [Background] Gill H, Kumana CR, Yim R, Hwang YY, Chan TSY, Yip SF, Lee HKK, Mak V, Lau JSM, Chan CC, Kho B, Wong RSM, Li W, Lin SY, Lau CK, Ip HW, Leung RYY, Lam CCK, Kwong YL. Oral arsenic trioxide incorporation into frontline treatment with all-trans retinoic acid and chemotherapy in newly diagnosed acute promyelocytic leukemia: A 5-year prospective study. Cancer. 2019 Sep 1;125(17):3001-3012. doi: 10.1002/cncr.32180. Epub 2019 May 15. PMID 31090936
- [Background] Gill HS, Yim R, Kumana CR, Tse E, Kwong YL. Oral arsenic trioxide, all-trans retinoic acid, and ascorbic acid maintenance after first complete remission in acute promyelocytic leukemia: Long-term results and unique prognostic indicators. Cancer. 2020 Jul 15;126(14):3244-3254. doi: 10.1002/cncr.32937. Epub 2020 May 4. PMID 32365228
- [Background] Kumana CR, Mak R, Kwong YL, Gill H. Resurrection of Oral Arsenic Trioxide for Treating Acute Promyelocytic Leukaemia: A Historical Account From Bedside to Bench to Bedside. Front Oncol. 2020 Aug 4;10:1294. doi: 10.3389/fonc.2020.01294. eCollection 2020. PMID 32850403